CLINICAL TRIAL: NCT06968780
Title: Buccal Pad of Fat Graft vs. Palatal Rotation Scarf Graft for Soft Tissue Enhancement and Prevention of Dehiscence Around Zygomatic Implants Placed in Patients With Severely Atrophic Maxilla: A Randomized Clinical Trial
Brief Title: Buccal Fat Pad vs. Palatal Rotation Scarf Grafts for Soft Tissue Management Around Zygomatic Implants
Acronym: RCT BFP ZAGA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Khaled Mohamed Allam, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ZYGO-RCT-BFPvsPRG-2025
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Zygomatic Implants; Atrophic Maxilla; Soft Tissue Defect; Soft Tissue Healing
Keywords: ZAGA; Zygomatic Implants; Buccal Fat Pad; BFP; Palatal Rotation Graft; PRG; Scarf Graft; Atrophic Maxilla; Soft tissue Recession; Dehiscence; RCT; Zygoma; Implant
MeSH Terms: conditions — Atrophic Maxilla | interventions — 2-benzyl-3-formylpropanoic acid

STUDY DESIGN:
Intervention Model Description: 1. Superiority test.
  2. Randomized Controlled Clinical Trial.
  3. Parallel group study.
  4. Allocation Ratio 1:1.
Who Masked: Participant, Outcomes Assessor
Masking Description: Each patient will be given a code by the researcher and the observers will be blind to which group this case belong. Patients, radiographic outcome assessor and statistician will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zygomatic implants placed using ZAGA approach & Buccal Fat Pad (Experimental): All patients involved in this study will be divided into two groups, each group will receive Zygomatic implants (Exteriorized ZAGA approach) alone (dual bilateral, quad) or in combination with axial implants if bone permits(hybrid). The first group (Control Group) will be treated with the buccal pad of fat graft, while the other (Study Group) is going to be treated by the palatal scarf graft after implant placement.
  BFP has a long successful history in oral surgery for its use in closure of Oroantral communication and taking advantage of the fact that it contains progenitor stem cells showing similar phenotype with (ASC) adipose-derived stem cells characteristics, which can similarly differentiate into the chondrogenic, adipogenic, or osteogenic lineage. Making them an invaluable reservoir for tissue engineering.
  Interventions: Procedure: Buccal Fat Pad
- Zygomatic implants placed using ZAGA approach & Palatal Rotation Scarf Graft (Experimental): All patients involved in this study will be divided into two groups, each group will receive Zygomatic implants (Exteriorized ZAGA approach) alone (dual bilateral, quad) or in combination with axial implants if bone permits(hybrid). The first group (Control Group) will be treated with the buccal pad of fat graft, while the other (Study Group) is going to be treated by the palatal scarf graft after implant placement.
  This technique uses tissue from the palatal area, which has a rich blood supply placed around the neck of the zygomatic implant aiming to protect the mucosal tissues buccal to the exteriorized implants from capillary compression and subsequent soft tissue recession. The palatal rotation scarf graft has been proven to provide a robust, resilient soft tissue flap with good potential for long-term stability and esthetic outcomes around implants
  Interventions: Procedure: Palatal Rotation Scarf Graft

INTERVENTIONS:
Procedure: Buccal Fat Pad — BFP has a long successful history in oral surgery for its use in closure of Oroantral communication and taking advantage of the fact that it contains progenitor stem cells showing similar phenotype with (ASC) adipose-derived stem cells characteristics, which can similarly differentiate into the chondrogenic, adipogenic, or osteogenic lineage. Making them an invaluable reservoir for tissue engineering.
  Other Names: Buccal pad of fat; BFP
  Arms: Zygomatic implants placed using ZAGA approach & Buccal Fat Pad
Procedure: Palatal Rotation Scarf Graft — This technique uses tissue from the palatal area, which has a rich blood supply placed around the neck of the zygomatic implant aiming to protect the mucosal tissues buccal to the exteriorized implants from capillary compression and subsequent soft tissue recession. The palatal rotation scarf graft has been proven to provide a robust, resilient soft tissue flap with good potential for long-term stability and esthetic outcomes around implants.
  Other Names: Scarf Graft; Palatal pedicled graft; Palatal graft flap
  Arms: Zygomatic implants placed using ZAGA approach & Palatal Rotation Scarf Graft

SUMMARY:
Over the past 20 years, the demand for oral rehabilitation among edentulous patients has steadily increased. Traditionally, individuals with edentulous maxillae were treated using removable complete dentures. However, these often result in poor patient satisfaction due to instability and functional limitations. Dental rehabilitation with implants in the maxillary arch presents unique challenges, primarily due to the anatomical complexity of the maxilla and the need for adequate residual ridge dimensions for successful implant placement.

Following the extraction of maxillary teeth, patients experience rapid and progressive alveolar bone loss in both vertical and horizontal dimensions. This resorption is largely attributed to the absence of teeth and periodontal ligament fibers support, which are essential for transmitting mechanical forces that maintain bone homeostasis. In addition, the loss of maxillary molars accelerates pneumatization/expansion of the maxillary sinus, further reducing available bone volume. Contributing factors such as ill-fitting dentures and systemic health conditions can exacerbate this process, complicating implant placement even further.

To overcome these limitations, oral and maxillofacial surgeons have developed a range of advanced techniques, including tilted implants, sinus floor elevation, short implants, pterygoid implants, and most notably, zygomatic implants. Zygomatic implants bypass the atrophic alveolar ridge entirely by anchoring into the dense zygomatic bone, offering a reliable solution for patients with severely resorbed maxillae who are not candidates for conventional implant therapy.

DETAILED DESCRIPTION:
The study aims to compare two different soft tissue augmentation techniques-buccal fat pad graft and palatal rotation scarf graft-to determine which method is more effective in enhancing soft tissue volume, improving tissue stability, and preventing dehiscence around zygomatic implants. Both grafts have shown promise in separate clinical applications, but this head-to-head comparison it will help in identifying the more optimal and predictable graft technique, the research aims to improve clinical outcomes, reduce complications, and enhance the long-term success of zygomatic implants in challenging clinical scenarios.

ELIGIBILITY:
Inclusion Criteria:

1. Patient of age 18 years or more, who can understand and sign an informed consent.
2. Patients with severely atrophic edentulous upper arch (Cawood & Howell class IV, V, VI) that could not be restored by standard axial implants without augmentation.
3. Patients with severely atrophic edentulous upper arch (Bedrossian classification inadequate bone in zones II or III or all three zones) that could not be restored by standard axial implants without augmentation.
4. Good systemic health (ASA score I-II)
5. Highly motivated patients with good compliance to oral hygiene habits.

Exclusion Criteria:

1. Patients with cardiovascular disease or pulmonary disease or medical systemic condition that does not permit the surgical procedure under general anesthesia (ASA III, IV, V and VI).
2. Patients with conditions contraindicating implant placement (e.g.: radiation to the head and neck, intra-venous bisphosphonates, uncontrolled Diabetes mellitus).
3. Heavy smokers. (> 20 cigarettes daily)
4. Patient with psychiatric problems, severe bruxism, or other parafunctional habits.
5. Acute maxillary sinus infection or untreated maxillary sinus cyst.
6. Malignancy or pathology in Maxilla or Zygoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Peri-implant Soft-Tissue Recessions (PSTR), Condition & Quality | 6 months
  Incidence of dehiscence and peri-implantitis based on clinical examination, reference photographs obtained, signs of infection, keratinized soft tissue thickness using periodontal probe.

SECONDARY OUTCOMES:
Implant Survival Rate | 6 months
  ORIS Success Criteria of Zygomatic Implants

CONTACTS AND LOCATIONS:
Overall Officials: Ramy R El-Beialy, PhD, Study Director — Cairo University
Locations (1):
- Cairo University, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Outcomes results
Supporting Information: Study Protocol, ICF, CSR

REFERENCES:
- [Background] Blanco-Ruiz S, Molinero-Mourelle P, Blanco-Ruiz M, Fernandez-Tresguerres FG, Blanco-Samper S, Lopez-Quiles J. Effect of the buccal fat pad in the prevention of zygomatic implant surgery postoperative complications: A pilot study. Med Oral Patol Oral Cir Bucal. 2023 Jul 1;28(4):e371-e377. doi: 10.4317/medoral.25792. PMID 37330966
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/37330966/